CLINICAL TRIAL: NCT02120261
Title: Using Saline for Myofascial Pain Syndromes (USAMPS)
Acronym: USAMPS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of activity, Primary researcher moved to another institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Carlos Roldan, Associate Professor of EMS, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-14-0072
Record Dates: First submitted 2014-04-14; First posted 2014-04-22 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Myofascial Pain Syndrome
Keywords: Myofascial Pain Syndrome; trigger point injection
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Saline Solution; Lidocaine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPI with Normal Saline (Experimental): Trigger point injection (TPI) with 1 mL of normal saline solution. Trigger point injection involves a single injection in the area of maximal tenderness or trigger point. This will be performed by the treating physician under sterile technique with a 25 gauge needle.
  Interventions: Drug: Normal Saline
- TPI with Lidocaine & Triamcinolone Acetonide (Active Comparator): Trigger point injection (TPI) with 1 mL of conventional drug mix (lidocaine 1%; 10 mL+ triamcinolone acetonide 40 mg/mL). Trigger point injection involves a single injection in the area of maximal tenderness or trigger point. This will be performed by the treating physician under sterile technique with a 25 gauge needle.
  Interventions: Drug: Lidocaine Hydrochloride; Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: Normal Saline — Trigger point injection (TPI) with 1 mL of normal saline solution. Trigger point injection involves a single injection in the area of maximal tenderness or trigger point. This will be performed by the treating physician under sterile technique with a 25 gauge needle.
  Arms: TPI with Normal Saline
Drug: Lidocaine Hydrochloride — Trigger point injection (TPI) with 1 mL of conventional drug mix (lidocaine 1%; 10 mL+ triamcinolone acetonide 40 mg/mL). Trigger point injection involves a single injection in the area of maximal tenderness or trigger point. This will be performed by the treating physician under sterile technique with a 25 gauge needle.
  Arms: TPI with Lidocaine & Triamcinolone Acetonide
Drug: Triamcinolone acetonide — Trigger point injection (TPI) with 1 mL of conventional drug mix (lidocaine 1%; 10 mL+ triamcinolone acetonide 40 mg/mL). Trigger point injection involves a single injection in the area of maximal tenderness or trigger point. This will be performed by the treating physician under sterile technique with a 25 gauge needle.
  Arms: TPI with Lidocaine & Triamcinolone Acetonide

SUMMARY:
This study involves adult patients diagnosed with Myofascial Pain Syndromes (MPS). The purpose of this research study is to determine if there is a therapeutic difference between trigger point injection (TPI) of normal saline and conventional drug mix (local anesthesic + steroid) in treating MPS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with MPS of the trapezius, gluteus medius/minimus, iliocostalis thoracis-lumborum, quadratus Lumborum, or paraspinal muscles in the emergency department.

Exclusion Criteria:

* Patients allergic to lidocaine and/or steroids.
* Pregnant women.
* Prisoners.
* Patients who are cognitively impaired and/or unable to consent for the study.
* Age < 18.
* Signs of localized infection or skin breakdown at the injection site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Roldan, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Memorial Hermann Hospital Texas Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants who were enrolled did not start the study.
Period: Overall Study
Arm/Group | TPI With Normal Saline | TPI With Lidocaine & Triamcinolone Acetonide
Started | 23 | 25
Completed | 23 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TPI With Normal Saline | TPI With Lidocaine & Triamcinolone Acetonide | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 25 | 48
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 12 | 13 | 25
  Race/Ethnicity: African American or Black | 8 | 8 | 16
  Race/Ethnicity: White | 3 | 3 | 6
  Race/Ethnicity: Asian | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: The level of pain intensity is quantified using a standard 0-10 Numerical Rating Scale with 10 being the most severe pain intensity and 0 the absence of pain.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TPI With Normal Saline | TPI With Lidocaine & Triamcinolone Acetonide
Number analyzed (Participants) | 23 | 25
units on a scale | 7.69 (1.87) | 7.44 (2.04)

2. Primary Outcome: Pain Intensity
Description: as for outcome 1
Time Frame: at discharge (a few minutes after receiving intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TPI With Normal Saline | TPI With Lidocaine & Triamcinolone Acetonide
Number analyzed (Participants) | 23 | 25
units on a scale | 1.52 (2.22) | 1.76 (2.86)

3. Primary Outcome: Pain Intensity
Description: as for outcome 1
Time Frame: 2 weeks
Population: Pain intensity was not measured in 6 subjects in the TPI with Normal Saline arm and 4 subjects in the TPI with Lidocaine & Triamcinolone Acetonide arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TPI With Normal Saline | TPI With Lidocaine & Triamcinolone Acetonide
Number analyzed (Participants) | 17 | 21
units on a scale | 4.29 (3.66) | 4.14 (3.17)

4. Secondary Outcome: Duration of Pain Relief
Description: If the patient experienced pain relief with the trigger point injection and the pain came back later, the number of days after the injection at which the pain had returned was recorded.
Time Frame: 16 days
Measure: Median (Full Range); unit: days
Arm/Group | TPI With Normal Saline | TPI With Lidocaine & Triamcinolone Acetonide
Number analyzed (Participants) | 23 | 25
days | 3 [1 to 16] | 1 [0 to 15]

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- TPI With Normal Saline: Trigger point injection (TPI) with 1 mL of normal saline solution. Trigger point injection involves a single injection in the area of maximal tenderness or trigger point.
  Normal Saline: Trigger point injection (TPI) with 1 mL of normal saline solution. Trigger point injection involves a single injection in the area of maximal tenderness or trigger point.
- TPI With Lidocaine & Triamcinolone Acetonide: Trigger point injection (TPI) with 1 mL of conventional drug mix (lidocaine 1%; 10 mL+ triamcinolone acetonide 40 mg/mL). Trigger point injection involves a single injection in the area of maximal tenderness or trigger point.
  Lidocaine Hydrochloride: Trigger point injection (TPI) with 1 mL of conventional drug mix (lidocaine 1%; 10 mL+ triamcinolone acetonide 40 mg/mL). Trigger point injection involves a single injection in the area of maximal tenderness or trigger point.
  Triamcinolone acetonide: Trigger point injection (TPI) with 1 mL of conventional drug mix (lidocaine 1%; 10 mL+ triamcinolone acetonide 40 mg/mL). Trigger point injection involves a single injection in the area of maximal tenderness or trigger point.
Arm/Group | TPI With Normal Saline | TPI With Lidocaine & Triamcinolone Acetonide
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes